CLINICAL TRIAL: NCT05304338
Title: Evaluation of the Effect of Oil Pulling on Dental and Gingival Health
Brief Title: Evaluation of the Effect of Oil Pulling
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Ahmet Bedreddin Şahin, Research assistant, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 8948
Record Dates: First submitted 2022-03-22; First posted 2022-03-31 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Oral Hygiene; Dental Plaque
Keywords: Chlorhexidine; Oil pulling; Plaque Regrowth model; Coconut oil; Digital spectrophotometer
MeSH Terms: conditions — Dental Plaque | interventions — Chlorhexidine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Chlorhexidine (Active Comparator)
  Interventions: Drug: Chlorhexidine
- Coconut Oil (Experimental)
  Interventions: Other: Oil Pulling
- Black Cumin Oil (Experimental)
  Interventions: Other: Oil Pulling
- Terebinth Oil (Experimental)
  Interventions: Other: Oil Pulling
- Distilled Water (Placebo Comparator)
  Interventions: Other: Distilled Water

INTERVENTIONS:
Drug: Chlorhexidine — Gargling with 10 mL 0.2% Chlorhexidine
  Arms: Chlorhexidine
Other: Oil Pulling — In oil pulling therapy, a tablespoon of edible oil is placed in the mouth and swirled between the teeth for 15 to 20 minutes
  Arms: Black Cumin Oil; Coconut Oil; Terebinth Oil
Other: Distilled Water — Gargling with 10 mL distilled water
  Arms: Distilled Water

SUMMARY:
The objectives of this study were to evaluate the inhibitory effect on plaque and the tooth discoloration associated with agents used in the chemical plaque control of oil pulling in comparison with chlorhexidine-containing mouthwash and water in a four-day plaque regrowth model.

One hundred dentistry students were included in this randomized, parallel-group, placebo-controlled clinical study. In this study, participants were divided into 5 equal groups: Group 1: Gargling with 0.2% chlorhexidine; Group 2: Oil pulling with coconut oil; Group 3: Oil pulling with black cumin oil; Group 4: Oil pulling with terebinth oil; Group 4: Gargling with distilled water. Participants were instructed to refrain from mechanical oral hygiene and rinse only with the allocated mouth rinse during the four-day period. The differences in plaque index, gingival index, and tooth discoloration were evaluated in the study.

ELIGIBILITY:
Inclusion Criteria:

* Without systemic disease,
* Had at least 24 teeth, and
* Without fixed or removable prostheses or orthodontic appliances

Exclusion Criteria:

* Individuals with a history of systemic or topical oral antimicrobial therapy use in the last 3 months
* Individuals with an allergy to any ingredient used in the study
* Smokers
* Pregnant or breastfeeding women
* Individuals with ≥2 mm gingival recession

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2021-10-10 (Actual); Primary Completion 2021-11-25 (Actual); Study Completion 2022-01-21 (Actual)

PRIMARY OUTCOMES:
Dental Plaque | Day 4
  Plaque scores recorded by using the Quigley-Hein and Turesky plaque index (Q-H).

SECONDARY OUTCOMES:
Tooth Color | Day 1- Day 4
  The tooth color was determined with a digital spectrophotometer

CONTACTS AND LOCATIONS:
Locations (1):
- Ataturk University, Erzurum, None Selected, Turkey (Türkiye)

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-09-01): https://cdn.clinicaltrials.gov/large-docs/38/NCT05304338/Prot_SAP_000.pdf
  • Informed Consent Form (2021-09-01): https://cdn.clinicaltrials.gov/large-docs/38/NCT05304338/ICF_001.pdf